CLINICAL TRIAL: NCT01075074
Title: The Effect of Pre Operative Transversus Abdominis Plane (TAP) Block in the Quality of Recovery of Patients Undergoing Outpatient Laparoscopic Gynecological Surgery: A Prospective, Randomized Blinded Study
Brief Title: Pre Operative Transversus Abdominis Plane Block Laparoscopic Gynecological Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Gildasio De Oliveira, Gildasio De Oliveira, M.D. Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STU00023475
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Results first posted 2012-04-03 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-10

CONDITIONS: Pain; Surgery
Keywords: Pain; TAP block; Laparoscopic; Gynecologic
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ropivacaine 0.05% (Active Comparator): Subject received a bilateral transversus abdominis plane block block using 15 cc of 0.5% ropivacaine on each side
  Interventions: Procedure: Transversus abdominis plane block
- Normal Saline (Placebo Comparator): Subjects received a bilateral transversus abdominis plane block using 15 cc of sterile normal saline.
  Interventions: Procedure: Transversus abdominis plane block
- Ropivacaine 0.25% (Active Comparator): Subjects received a bilateral transversus abdominis plane block using 15cc of 0.25% ropivacaine on each side
  Interventions: Procedure: Transversus abdominis plane block

INTERVENTIONS:
Procedure: Transversus abdominis plane block — A regional block performed in the transversus abdominis plane of the abdomen, used to provide anesthesia and analgesia for the abdominal region.
  Other Names: TAP block

SUMMARY:
The use of pre-operative transversus abdominis plane block will reduce pain after outpatient laparoscopic gynecological surgery and improve quality of recovery.

DETAILED DESCRIPTION:
75 subjects will be randomly allocated into 3 groups, using a computer generated table of random numbers. Group A (study group) will receive a bilateral TAP block using 15 cc of 0.5% ropivacaine on each side. Group B (control group) will receive 15 cc of sterile normal saline. Group C (study group 2) will receive a bilateral TAP block using 15 cc of 0.25% ropivacaine on each side.

Subjects will be premedicated with intravenous (IV) midazolam 0.04 mg/kg. Routine ASA monitors will be applied. Anesthesia will be induced with remifentanil infusion started at 0.1 mcg/kg/minute titrated to keep blood pressure within 20% of the baseline and propofol 1.0 -2.0 mg/kg. Tracheal intubation will be facilitated with rocuronium (0.6 mg/kg) or succinylcholine (1-2mg /kg). After induction, a bilateral TAP block will be performed in both groups, under ultrasound guidance with a transportable ultrasound device (SonoSite, Bothell, WA, USA) and a linear 6-13 MHz ultrasound transducer .Once the EOAM, IOAM and TAM are visualized at the level of the anterior axillary line between the 12th rib and the iliac crest, the puncture area and the ultrasound probe will be prepared in a sterile manner. Then the block will be performed with a 21 G 90mm StimuQuik needle( Arrow International, Reading, PA, USA ) utilizing an "in- plane" ultrasound-guided technique by three investigators (GDO ,AP). Once the tip of the needle is placed in the space between the IOAM and TAM, and after negative aspiration of blood, 15 cc of 0.5% ropivacaine, 15 cc of 0.25% ropivacaine or sterile normal saline will be administered under direct ultrasonographic guidance. The contralateral block will be performed in the same fashion. Anesthesia will be maintained with sevoflurane titrated to maintain a bispectral index (BIS) between 40-60 , remifentanil infusion started at 0.1mcg/kg/min titrated to keep blood pressure within 20 % of baseline values , and rocuronium that will be administered at the discretion of the anesthesiologist. Upon termination of the surgery, neuromuscular blockade will be antagonized with a combination of neostigmine 0.05mg/kg and glycopyrrolate 0.01 mg/kg. Subjects will also receive ketorolac 30 mg IV after discontinuation of remifentanil for postoperative pain control. Ondansetron 4 mg IV will be administered to prevent postoperative nausea and vomiting. Subjects will be assessed in the OR after extubation for their pain using a numerical rating scale and if pain greater than 4/10 they will receive hydromorphone(10 mcg /kg IV) Subjects will receive IV Hydromorphone in divided doses as needed to achieve a verbal rating score for pain <4 out of 10 In PACU.They will also receive metoclopramide (20 mg IV ) as rescue antiemetic in PACU. The primary and secondary outcomes will be assessed by an independent observer who will be blinded to group allocation (CA, AP, SA, YV, RJM and PF). A study team representative will telephone the participant at 24 hours, to complete the modified quality of recovery (QOR40) survey and ask the following:

1. How much pain they are experiencing 0-10
2. How and what kind of pain medications have been used since discharge.
3. If they have had any nausea
4. What kind of nausea relief medications have been used since discharge

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-64 years
* Surgery: Outpatient Gynecological laparoscopic surgery
* ASA status: I and II
* Fluent in English

Exclusion Criteria:

* History of allergy to local anesthetics
* History of chronic opioid use
* Pregnant patients
* BMI greater than 30

Drop-out criteria:

* Patient or surgeon request
* Complications related to the procedure

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2010-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gildasio DeOliveira, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Lovatsis D, Jose JB, Tufman A, Drutz HP, Murphy K. Assessment of patient satisfaction with postoperative pain management after ambulatory gynaecologic laparoscopy. J Obstet Gynaecol Can. 2007 Aug;29(8):664-7. doi: 10.1016/s1701-2163(16)32552-x. PMID 17714620
- [Background] Wills VL, Hunt DR. Pain after laparoscopic cholecystectomy. Br J Surg. 2000 Mar;87(3):273-84. doi: 10.1046/j.1365-2168.2000.01374.x. PMID 10718794
- [Background] Goldstein A, Grimault P, Henique A, Keller M, Fortin A, Darai E. Preventing postoperative pain by local anesthetic instillation after laparoscopic gynecologic surgery: a placebo-controlled comparison of bupivacaine and ropivacaine. Anesth Analg. 2000 Aug;91(2):403-7. doi: 10.1097/00000539-200008000-00032. PMID 10910857
- [Background] Shaw IC, Stevens J, Krishnamurthy S. The influence of intraperitoneal bupivacaine on pain following major laparoscopic gynaecological procedures. Anaesthesia. 2001 Nov;56(11):1041-4. doi: 10.1046/j.1365-2044.2001.02215.x. PMID 11703235
- [Background] Moiniche S, Mikkelsen S, Wetterslev J, Dahl JB. A qualitative systematic review of incisional local anaesthesia for postoperative pain relief after abdominal operations. Br J Anaesth. 1998 Sep;81(3):377-83. doi: 10.1093/bja/81.3.377. PMID 9861124
- [Background] Keita H, Benifla JL, Le Bouar V, Porcher R, Wachowska B, Bedairia K, Mantz J, Desmonts JM. Prophylactic ip injection of bupivacaine and/or morphine does not improve postoperative analgesia after laparoscopic gynecologic surgery. Can J Anaesth. 2003 Apr;50(4):362-7. doi: 10.1007/BF03021033. PMID 12670813
- [Background] Buvanendran A, Kroin JS. Multimodal analgesia for controlling acute postoperative pain. Curr Opin Anaesthesiol. 2009 Oct;22(5):588-93. doi: 10.1097/ACO.0b013e328330373a. PMID 19606021
- [Background] Turner GA, Chalkiadis G. Comparison of preoperative with postoperative lignocaine infiltration on postoperative analgesic requirements. Br J Anaesth. 1994 May;72(5):541-3. doi: 10.1093/bja/72.5.541. PMID 8198905
- [Background] O'Donnell BD, McDonnell JG, McShane AJ. The transversus abdominis plane (TAP) block in open retropubic prostatectomy. Reg Anesth Pain Med. 2006 Jan-Feb;31(1):91. doi: 10.1016/j.rapm.2005.10.006. No abstract available. PMID 16418039
- [Background] Hebbard P, Fujiwara Y, Shibata Y, Royse C. Ultrasound-guided transversus abdominis plane (TAP) block. Anaesth Intensive Care. 2007 Aug;35(4):616-7. No abstract available. PMID 18020088

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from Prentice Women's Hospital consecutively from 04/01/2010-02/2011
Groups:
- Ropivacaine 0.05%: Subjects received a bilateral transversus abdominis plane block block using 15 cc of 0.5% ropivacaine
- Normal Saline: Subjects received a transversus abdominis plane block using 15 cc of sterile normal saline
- Ropivacaine 0.25%: Subjects received a bilateral transversus abdominis plane block using 15cc of ropivacaine 0.025%
Period: Overall Study
Arm/Group | Ropivacaine 0.05% | Normal Saline | Ropivacaine 0.25%
Started | 25 | 25 | 25
Completed | 24 | 23 | 23
Not Completed | 1 | 2 | 2
Not completed — Surgeon changed to open incisional case | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ropivacaine 0.05% | Normal Saline | Ropivacaine 0.25% | Total
Number analyzed (Participants) | 25 | 25 | 25 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 25 | 75
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 38 (8) | 38 (10) | 35 (9) | 37 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 25 | 75
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 25 | 75

OUTCOME MEASURES:

1. Primary Outcome: The Quality of Recovery Questionnaire (QoR40) on the Day (24 Hours) After Surgery
Description: The quality of recovery questionnaire (QOR40) is a 40 question assessment of patient recovery following surgery. It evaluates 5 domains of recovery: pain, emotional status, physical comfort, physical independence, and support. Each question is scores on a 1 to 5 Likert scale with total scores ranging for 40, representing poor recovery, to 200, representing outstanding recovery.
Time Frame: 24 hours after surgery
Population: 75 subjects were randomized in 3 groups of 25, 5 were excluded from analysis because the surgeon had to proceed to an open incision from a laparoscopic case during the procedure.
Measure: Median (Full Range); unit: units on a scale
Groups:
- Ropivacaine 0.5%: The ropivacaine 0.5% group will receive a bilateral transversus abdominal plane block using 15 cc of 0.5% ropivacaine on each side
- Normal Saline: The control group will receive a bilateral transversus abdominal plane block using 15 cc of sterile normal saline.
- Ropivacaine 0.25%: The ropivacaine 0.25% group will receive a bilateral transversus abdominal plane block using 15 cc of 0.25% ropivacaine on each side
Arm/Group | Ropivacaine 0.5% | Normal Saline | Ropivacaine 0.25%
Number analyzed (Participants) | 24 | 23 | 23
units on a scale | 172 [160 to 190] | 157 [148 to 169] | 173 [165 to 189]
Statistical Analysis 1: Comparison: Ropivacaine 0.5% vs Normal Saline vs Ropivacaine 0.25%; A sample size of 23 subjects per group was estimated to achieve 80% power to detect a 10 point difference in the aggregated QOR40 score for the 3 study groups to be compared assuming an overall standard deviation of 12; Test type: Superiority or Other; p = 0.006, Kruskal-Wallis — Corrected for 6 comparisons
Statistical Analysis 2: Comparison: Ropivacaine 0.5% vs Normal Saline; Test type: Superiority or Other; p = 0.03, Wilcoxon (Mann-Whitney); Median Difference (Net) = 16, 95% CI 2-sided [1 to 30]
Statistical Analysis 3: Comparison: Normal Saline vs Ropivacaine 0.25%; Test type: Superiority or Other; p = 0.01, Wilcoxon (Mann-Whitney); Median Difference (Net) = 17, 95% CI 2-sided [2 to 31]
Statistical Analysis 4: Comparison: Ropivacaine 0.5% vs Ropivacaine 0.25%; Test type: Superiority or Other; p = 1.0, Wilcoxon (Mann-Whitney); Median Difference (Net) = 1, 95% CI 2-sided [-16 to 12]

2. Secondary Outcome: Pain Burden During Early Recovery From Anesthesia
Description: Area under the numeric rating scale for pain versus time (min) curve during the post anesthesia care admission. Numeric rating scale 0 to 10 with 0 equals no pain and 10 equals worst pain imaginable.
Time Frame: Post Operative
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale * minutes
Groups:
- Normal Saline: The normal saline group will receive a bilateral transversus abdominal plane block using 15 cc of sterile normal saline.
Arm/Group | Ropivacaine 0.5% | Normal Saline | Ropivacaine 0.25%
Number analyzed (Participants) | 24 | 23 | 23
score on a scale * minutes | 210 (4) [90 to 345] | 405 (4) [360 to 502] | 210 (4) [135 to 365]
Statistical Analysis 1: Comparison: Ropivacaine 0.5% vs Normal Saline vs Ropivacaine 0.25%; Test type: Superiority or Other; p = 0.0003, Kruskal-Wallis — P values is corrected for 6 comparisons
Statistical Analysis 2: Comparison: Ropivacaine 0.5% vs Normal Saline vs Ropivacaine 0.25%; Test type: Superiority or Other; p = 0.0003, Kruskal-Wallis — Corrected for 6 comparisons
Statistical Analysis 3: Comparison: Ropivacaine 0.5% vs Normal Saline; Test type: Superiority or Other; p = 0.0004, Wilcoxon (Mann-Whitney); Median Difference (Net) = 195, 95% CI 2-sided [98 to 300]
Statistical Analysis 4: Comparison: Normal Saline vs Ropivacaine 0.25%; Test type: Superiority or Other; p = 0.0003, Wilcoxon (Mann-Whitney); Median Difference (Net) = 195, 95% CI 2-sided [98 to 278]
Statistical Analysis 5: Comparison: Ropivacaine 0.5% vs Ropivacaine 0.25%; Test type: Superiority or Other; p = 0.86, Wilcoxon (Mann-Whitney); Median Difference (Net) = 0, 95% CI 2-sided [-105 to 83]

3. Secondary Outcome: Opioid Pain Medications Consumed During the First 24 Hours Post Surgery
Description: Opioid consumption in oral morphine equivalents taken by the subject for pain during the first 24 hours post hospital discharge
Time Frame: 24 hours
Population: as for outcome 1
Measure: Mean (Full Range); unit: mEq of PO morphine equivalent
Groups:
- Ropivacaine 0.5%: Ropivacaine 0.5% group will receive a bilateral transversus abdominis plane block block using 15 cc of 0.5% ropivacaine on each side
- Normal Saline: Normal saline group will receive a bilateral transversus abdominis plane block 15 cc of sterile normal saline.
- Ropivacaine 0.25%: Ropivicaine 0.25% group will receive a bilateral transversus abdominis plane block using 15 cc of 0.25% ropivacaine on each side
Arm/Group | Ropivacaine 0.5% | Normal Saline | Ropivacaine 0.25%
Number analyzed (Participants) | 21 | 23 | 22
mEq of PO morphine equivalent | 40 [13 to 72] | 78 [61 to 90] | 39 [25 to 58]
Statistical Analysis 1: Comparison: Ropivacaine 0.5% vs Normal Saline vs Ropivacaine 0.25%; Test type: Superiority or Other; p = 0.0005, Kruskal-Wallis — Corrected for multiple comparisons (n=6)
Statistical Analysis 2: Comparison: Ropivacaine 0.5% vs Normal Saline; Test type: Superiority or Other; p = 0.01, Wilcoxon (Mann-Whitney); Median Difference (Net) = 38, 95% CI 2-sided [8 to 50]
Statistical Analysis 3: Comparison: Normal Saline vs Ropivacaine 0.25%; Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney); Median Difference (Net) = 40, 95% CI 2-sided [12 to 47]
Statistical Analysis 4: Comparison: Ropivacaine 0.5% vs Ropivacaine 0.25%; Test type: Superiority or Other; p = 0.95, Wilcoxon (Mann-Whitney); Median Difference (Net) = 1, 95% CI 2-sided [-18 to 20]

4. Secondary Outcome: Time to Hospital Discharge Readiness
Description: Elapsed time from post anesthesia care unit to readiness to hospital discharge. Assessment were made using the modified post anesthetic discharge scoring system. This assess 5 criteria: vital signs, activity and mental status, pain nausea and/or vomiting, surgical bleed, and intake and output. A score greater than or equal to 9 (on a 0 to 10 scale) is considered ready for discharge.
Time Frame: 24 hours
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Ropivacaine 0.5% | Normal Saline | Ropivacaine 0.25%
Number analyzed (Participants) | 24 | 23 | 23
minutes | 90 [75 to 120] | 120 [105 to 150] | 90 [75 to 135]
Statistical Analysis 1: Comparison: Ropivacaine 0.5% vs Normal Saline; Test type: Superiority or Other; p = 0.03, Kruskal-Wallis — Corrected for multiple comparisons (n=6)
Statistical Analysis 2: Comparison: Ropivacaine 0.5% vs Normal Saline; Test type: Superiority or Other; p = 0.01, Wilcoxon (Mann-Whitney); Median Difference (Net) = 30, 95% CI 2-sided [0 to 60]
Statistical Analysis 3: Comparison: Normal Saline vs Ropivacaine 0.25%; Test type: Superiority or Other; p = 0.04, Wilcoxon (Mann-Whitney); Median Difference (Net) = 30, 95% CI 2-sided [0 to 60]
Statistical Analysis 4: Comparison: Ropivacaine 0.5% vs Ropivacaine 0.25%; Test type: Superiority or Other; p = 0.92, Wilcoxon (Mann-Whitney); Median Difference (Net) = 0, 95% CI 2-sided [-30 to 30]

ADVERSE EVENTS:
Time Frame: Post anesthesia care unit until discharge
Groups:
- Ropivacaine 0.5%: Subjects received a bilateral transversus abdominis plane block using 15 cc of 0.5% ropivacaine
- Ropivacaine 0.25%: Subjects received a bilateral transversus abdominis plane block using 15cc of ropivicaine 0.25%
Arm/Group | Ropivacaine 0.5% | Normal Saline | Ropivacaine 0.25%
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 12/25 | 11/25 | 12/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Ropivacaine 0.5% (N=25) | Normal Saline (N=25) | Ropivacaine 0.25% (N=25)
Nausea (Gastrointestinal disorders) | 12/24 (12) | 11/23 (11) | 12/23 (12)

LIMITATIONS AND CAVEATS:
We did not obtain local anesthetic levels to compare safety profile. We were underpowered to detect a difference in the physical comfort dimension of the QOR questionnaire between the ropivacaine groups and the saline group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes